CLINICAL TRIAL: NCT04588948
Title: A Pharmacokinetic Study of Intravitreal Aflibercept Injection in Vitrectomized and Non-vitrectomized Eyes With Diabetic Macular Edema
Acronym: DRAW-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not proceed due to funding issues.
Sponsor: Stanford University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Diana Do, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58689; VGFTe-DME-2041 (Other: Regeneron)
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: The study is an exploratory investigation to evaluate the intraocular and systemic pharmacokinetics of intravitreal aflibercept. A sample size of 60 eyes was chosen to provide a sample of 30 non-vitrectomized eyes and 30 vitrectomized eyes to evaluate. This sample size will allow for an initial determination of the pharmacokinetics of intravitreal aflibercept injection inside the eye and in the systemic circulation of eyes with DME.One eye per patient may be eligible. In this research proposal, participants will be followed for 12-month period and have 17 study visits
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitrectomized Eyes (Experimental): The study is an exploratory investigation to evaluate the intraocular and systemic pharmacokinetics of intravitreal aflibercept. A sample size of 60 eyes was chosen to provide a sample of 30 non-vitrectomized eyes and 30 vitrectomized eyes to evaluate.
  Interventions: Drug: Intravitreal Aflibercept
- Non-Vitrectomized Eyes (Experimental): The study is an exploratory investigation to evaluate the intraocular and systemic pharmacokinetics of intravitreal aflibercept. A sample size of 60 eyes was chosen to provide a sample of 30 non-vitrectomized eyes and 30 vitrectomized eyes to evaluate.
  Interventions: Drug: Intravitreal Aflibercept

INTERVENTIONS:
Drug: Intravitreal Aflibercept — Two arms (non-vitrectomized, and vitrectomized) are included in the study to evaluate the effect of vitrectomy on the intraocular and systemic pharmacokinetics of intravitreal aflibercept injection
  Other Names: Eylea

SUMMARY:
The primary objective is to investigate and characterize the intraocular pharmacokinetics (free and bound) following intravitreal aflibercept injection (IAI) in vitrectomized and non-vitrectomized eyes with diabetic macular edema

The secondary objectives are to -

* Investigate and characterize plasma concentrations (free and bound) following injections of intravitreal aflibercept in vitrectomized and non-vitrectomized eyes with diabetic macular edema
* Correlate with changes in ocular concentration of drug over 12 months -

  * change in Best Corrected Visual Acuity (BCVA)
  * change in Central Retinal Thickness (CRT)
  * change in Diabetic Retinopathy Severity Scale (DRSS)
  * changes observed on Ocular coherence tomography angiography (OCT-A)
  * number of injections
* Evaluate ocular and systemic safety of intravitreal aflibercept
* Additional plasma and anterior chamber (AC) fluid cytokine analysis will be performed if sufficient samples are available

DETAILED DESCRIPTION:
Little information is known about the intraocular pharmacokinetics of intravitreal aflibercept injection in human eyes of Diabetic macular edema (DME) patients. In addition, the durability of intravitreal aflibercept injection in vitrectomized eyes is not known, since individuals with a history of vitrectomy have been excluded from clinical trials in DME. Although we recently conducted a prospective study (the DRAW study) to evaluate the intraocular pharmacokinetics of IAI in eyes with neovascular age-related macular degeneration (AMD), this research did not include eyes with DME. There has been a paucity of studies on systemic levels of free aflibercept following intravitreal aflibercept injection in DME patients, which would have implications for normal vascular hemostasis and wound repair in which vascular endothelial growth factor (VEGF) plays an important role. The proposed research will fill in these gaps in the knowledge base for intravitreal aflibercept injection.

Two arms (non-vitrectomized, and vitrectomized) are included in the study to evaluate the effect of vitrectomy on the intraocular and systemic pharmacokinetics of intravitreal aflibercept injection. A sample size of 60 eyes was chosen to provide a sample of 30 non-vitrectomized eyes and 30 vitrectomized eyes to evaluate. This sample size will allow for an initial determination of the pharmacokinetics of intravitreal aflibercept injection inside the eye and in the systemic circulation of eyes with DME.

One eye per patient may be eligible. In this research proposal, participants will be followed for 12-month period. Study eyes will receive intravitreal aflibercept at baseline and then starting at month 2 there will be no mandatory injection. Subject will receive additional aflibercept on an as needed basis (PRN) if DME is still present. AC fluid and blood draw will be performed prior to first PRN dose of intravitreal aflibercept.

Study will involve following procedures: bio-microscopy, dilated fundoscopic exam, measurement of intraocular pressure, measurement of best corrected visual acuity (BCVA), fundus photograph, optical coherence tomography (OCT) and OCT-Angiography (OCT-A). Patients will be followed monthly for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* A patient must meet the following criteria to be eligible for inclusion in the study:

  * Age > 18 years with diabetes
  * Diabetic macular edema (DME) with
* 30 patients with non-vitrectomized eyes
* 30 patients with vitrectomized eyes

  • Prior DME treatment allowed if
* Intravitreal anti-VEGF agent 6 months before study day 0
* Intravitreal steroid administered 5 months before study day 0
* Laser photocoagulation administered 4 months before study day 0

  * Phakic and pseudophakic eyes are allowed in the study.
  * Willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures
  * Willing and able to comply with clinic visits and study-related procedures

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Presence of other retinal vascular diseases (AMD, vein occlusion) that could affect the VEGF levels within the eye
* History of fluocinolone acetonide intravitreal implant
* Known hypersensitivity to aflibercept
* Autoimmune disease of the anterior segment or posterior chamber including chronic keratoconjunctivitis sicca, uveitis, iritis/scleritis, blepharitis of either eye
* Infectious conjunctivitis, keratitis, or endophthalmitis of either eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0
* Any clinically significant acute or chronic medical condition that would preclude participation in a clinical study
* Pregnant or breastfeeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception prior to the initial dose/start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

  * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Intravitreal Aflibercept Pharmacokinetics | 12 months
  Intraocular aflibercept levels (free and bound) after intravitreal aflibercept injection.The primary objective is to investigate and characterize the intraocular pharmacokinetics (free and bound) following intravitreal aflibercept injection (IAI) in vitrectomized and non-vitrectomized eyes with diabetic macular edema

SECONDARY OUTCOMES:
Plasma aflibercept levels | 12 months
  • Investigate and characterize plasma concentrations (free and bound) following injections of intravitreal aflibercept in vitrectomized and non-vitrectomized eyes with diabetic macular edema
Correlation of drug concentration with ophthalmic outcomes | over 12 months
  Correlate with changes in ocular concentration of drug
  * change in BCVA
  * change in CRT
  * change in DRSS
  * changes observed on OCT-A
  * number of injections
Safety Outcomes | 12 months
  Compare adverse events during the trial to the expected adverse events on the Aflibercept label to assess ocular and systemic safety of intravitreal aflibercept.

CONTACTS AND LOCATIONS:
Overall Officials: David Brown, MD, Principal Investigator — Retina Consultants Houston
Locations (1):
- Byers Eye Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Hinai AS. Experience of intravitreal injections in a tertiary Hospital in Oman. Oman J Ophthalmol. 2015 Sep-Dec;8(3):166-70. doi: 10.4103/0974-620X.169896. PMID 26903722
- [Background] Semeraro F, Morescalchi F, Duse S, Parmeggiani F, Gambicorti E, Costagliola C. Aflibercept in wet AMD: specific role and optimal use. Drug Des Devel Ther. 2013 Aug 5;7:711-22. doi: 10.2147/DDDT.S40215. eCollection 2013. PMID 23990705
- [Background] Garcia-Quintanilla L, Luaces-Rodriguez A, Gil-Martinez M, Mondelo-Garcia C, Maronas O, Mangas-Sanjuan V, Gonzalez-Barcia M, Zarra-Ferro I, Aguiar P, Otero-Espinar FJ, Fernandez-Ferreiro A. Pharmacokinetics of Intravitreal Anti-VEGF Drugs in Age-Related Macular Degeneration. Pharmaceutics. 2019 Jul 31;11(8):365. doi: 10.3390/pharmaceutics11080365. PMID 31370346
- [Background] Kakinoki M, Sawada O, Sawada T, Saishin Y, Kawamura H, Ohji M. Effect of vitrectomy on aqueous VEGF concentration and pharmacokinetics of bevacizumab in macaque monkeys. Invest Ophthalmol Vis Sci. 2012 Aug 24;53(9):5877-80. doi: 10.1167/iovs.12-10164. PMID 22836776
- [Background] Ahn SJ, Ahn J, Park S, Kim H, Hwang DJ, Park JH, Park JY, Chung JY, Park KH, Woo SJ. Erratum. Intraocular Pharmacokinetics of Ranibizumab in Vitrectomized Versus Nonvitrectomized Eyes. Invest Ophthalmol Vis Sci. 2015 Mar 3;56(3):1473-4. doi: 10.1167/iovs.13-13054a. No abstract available. PMID 25737148